CLINICAL TRIAL: NCT06158659
Title: Improved Immunology Outcomes Associated With Feihe Lactoferrin Fortified With HMO in Infant Formula: A Randomized, Controlled Trial
Brief Title: Improved Immunology Outcomes Associated With Lactoferrin Fortified With HMO in Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 22-SM-11-FEIHE-002
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Flu; Cold
Keywords: infant formula; lactoferrin; HMO (Human Milk Oligosaccharides); immunology
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two arms of participants will be assigned masked products (investigational formula and control formula) after randomization, while the participants of breastfeeding arm will not be assigned study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feihe Investigational Formula (Experimental): Feihe Investigational Formula
  1. With the highest lactoferrin content (more than blue)
  2. Contains 2 kinds of HMOs
  3. Double probiotic combination
  4. Comprehensive nutrition: OPO, DHA&ARA, CPP, nucleotide, choline, inositol, taurine, L-carnitine, GOS, lutein
  Interventions: Dietary Supplement: Feihe Investigational Formula
- Control Formula (Active Comparator): Control formula contains comparable macronutrients and micronutrients, but does not contain Lactoferrin fortified with HMO
  Interventions: Dietary Supplement: Control Formula
- Breastfeeding (Other): breastmilk-feeding
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Dietary Supplement: Feihe Investigational Formula — Participants in this arm will receive stage 1 and stage 2 Feihe investigational formulas. At the first (up to) 6 months, they will be fed with stage1 formula, and then switch to stage 2 formula until 12 months.
  Arms: Feihe Investigational Formula
Dietary Supplement: Control Formula — Participants in this arm will receive stage 1 and stage 2 Control formulas. At the first (up to) 6 months, they will be fed with stage1 formula, and then switch to stage 2 formula until 12 months.
  Arms: Control Formula
Other: Breastfeeding — Exclusively breastfed for the first 4 months and continue with supplement food without any marketed infant formula.
  Arms: Breastfeeding

SUMMARY:
The goal of this interventional clinical trial is to test the effectiveness of enhancing immunity in newly born infants fed with Feihe investigational formula product containing Lactoferrin fortified with HMO. The main question it aims to answer is:

- whether the immunity functions of participants in terms of frequency of catching flu and cold in the study product arm is significantly better than participants assigned in the other two arms.

240 qualified participants will be randomized to 3 arms (investigational formula, control formula, and breast-feeding) to consume assigned formula or breast-feeding for 12 months according to protocol. There will be up to 6 site visits arranged for each participant during the study, and all relevant clinical and questionnaire data, including the most important primary outcome - frequency of catching flu and cold for each visit interval, will be captured, recorded and entered to CMTS (Clinical Management Trial System) for statistical analysis and reporting.

Researchers will compare the three arms to validate the assumption that the consumption of Feihe investigational formula product containing Lactoferrin fortified with HMO will improve immunity in newly born infants, along with physical development.

ELIGIBILITY:
Inclusion Criteria:

* Newborn baby, study entry before weaning (within 28 days of birth)
* Exclusively formula fed for at least 3 days prior to study entry and plan to be exclusively formula fed during the study (formula groups) OR plan to be exclusively fed with human milk during the study (breastfeeding group).
* Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age).
* Birth weight of 2500g (5 lbs. 8 oz.) to 4200g (9 lbs. 4 oz.).
* Signed informed consent obtained for infant's participation in the study.
* Parent or guardian of the infant agrees to not enroll the infant in another interventional clinical research study while participating in this study.

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant.
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion).
* Evidence of growth problems or concern for growth.
* Infant was born large for gestational age (LGA) (defined as birth weight-for-age exceeding 90th percentile as plotted on the growth chart provided by Feihe) from mother who was diabetic at childbirth.
* Participant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury.
* Use of probiotics/prebiotics before the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Frequency of flu and cold during the study | At the age of 12 months
  Frequency of flu and cold that participants caught during the study, which has positive relationship with immunology outcomes.

SECONDARY OUTCOMES:
Weight in grams | At the age of 15-28 days and 3, 6, 9, 12 months]
  The weight measurement (gram) of the participant for each site visit
Height in cm | At the age of 15-28 days and 3, 6, 9, 12 months
  The height measurement (cm) of the participant for each site visit
Head circumference in cm | At the age of 15-28 days and 3, 6, 9, 12 months
  The head circumference measurement (cm) of the participant for each site visit
Amount of formula intake in ml | At the age of 15-28 days and 3, 6, 9, 12 months
  The 24-Hour dietary recall of Formula intake (amount in ml of study formula, any other infant formula or milk consumed) of the participant for each site visit
Stool Characteristics Questionnaire | At the age of 15-28 days and 3, 6 months
  The frequency of bowel movements and the rating score (0-5) of the stool consistency over the 24-hour period. The rating score of the stool consistency from the stool picture:
  0-No bowel movement;
  1. Hard- dry, hard pellets;
  2. Formed- definite shape, not dry;
  3. Soft-no definite shape, pasty;
  4. Unformed or seedy- no shape, some water or small lumps ;
  5. Waterly- no shape, mainly water where the score of 0-1 represents poor stool characteristics, while 2-5 represents fine stool characteristics.
Medically-confirmed adverse events | baseline day to 12 months
  The frequency of medically-confirmed adverse events occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Zhang, MD, Principal Investigator — China National Center for Food Safety Risk Assessment Beijing, China
Locations (3):
- China (3):
  - Jinhua Nanyuan Community Health Center, Jinhua, Zhejiang
  - Li Pu Community Hospital, Jinhua, Zhejiang
  - Qiu Bin Community Hospital, Jinhua, Zhejiang